CLINICAL TRIAL: NCT03691207
Title: A Phase 2, Open-Label, Multi-center Study of AL101 in Patients With Adenoid Cystic Carcinoma (ACC) Bearing Activating Notch Mutations
Brief Title: A Study Of AL101In Patients With Adenoid Cystic Carcinoma (ACC) Bearing Activating Notch Mutations
Acronym: ACCURACY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ayala Pharmaceuticals, Inc, (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL-ACC-01
Record Dates: First submitted 2018-09-22; First posted 2018-10-01 (Actual); Results first posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Adenoid Cystic Carcinoma
MeSH Terms: conditions — Carcinoma, Adenoid Cystic

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SINGLE-ARM (Experimental): AL101 is an inhibitor of gamma secretase-mediated Notch signaling.
  Interventions: Drug: AL101

INTERVENTIONS:
Drug: AL101 — AL101 is a small-molecule that inhibits gamma secretase, an enzyme which plays a key role in the activation of the Notch signaling pathway by releasing the Notch intracellular domain (NICD) of all four Notch receptors from the membrane.
  In patients with aberrant Notch signaling, AL101 may inhibit Notch signaling and potentially impede tumor growth.The drug is administered intravenously
  Other Names: BMS 906024

SUMMARY:
This is a Phase 2, non comparative, open label, multicenter study of AL101 in patients with recurrent or metastatic ACC who harbor NOTCH 1,2,3,4 activating mutations.

DETAILED DESCRIPTION:
This is a Phase 2, non-comparative, open-label, multicenter study of AL101 in patients with recurrent or metastatic ACC who harbor NOTCH 1,2,3,4 activating mutations.

The study includes 2 cohorts, ran in a sequential fashion:

Cohort 1 - AL101 4 mg once weekly (QW) intravenously (IV) Cohort 2 - AL101 6 mg QW IV

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed Adenoid Cystic Carcinoma with known NOTCH 1/2/3/4 activating mutation that is recurrent or metastatic, not amenable to potentially curative surgery or radiotherapy.
2. Evidence of radiographic or clinical disease progression within 6-months of signing informed consent; newly diagnosed metastatic patients will be allowed.
3. Patients must have Formalin-fixed, Paraffin-embedded tissue available .
4. Must have at least 1 target lesion that is measurable for patients with nodal or visceral metastasis.

Exclusion Criteria:

1. Diagnosed with a malignancy other than ACC in the past 2 years.
2. Uncontrolled, Active Infection
3. Gastrointestinal (GI) disease with increased risk of diarrhea [e.g. inflammatory bowel disease (IBD)]
4. Symptomatic central nervous system (CNS) metastases.
5. Unstable or severe uncontrolled medical condition
6. Eastern Cooperative Oncology Group (ECOG) performance status ≥2.
7. Abnormal organ and marrow function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-12-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (10):
  - USC Norris Comprehensive Cancer center, Los Angeles, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic Hospital, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Canada (3):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Hamilton Health Sciences Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Center, London, Ontario
- Institut Gustave Roussy, Villejuif, France
- Rabin Medical center, Petah Tikva, Israel
- Radboud University, Nijmegen, Netherlands
- The Christie NHS Foundation Trust, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - AL101 4mg: AL101 4 mg once weekly (QW) intravenously (IV)
- Cohort 2 - AL101 6mg: AL101 6 mg once weekly (QW) intravenously (IV)
Period: Overall Study
Arm/Group | Cohort 1 - AL101 4mg | Cohort 2 - AL101 6mg
Started | 45 | 42
Completed | 0 | 0
Not Completed | 45 | 42
Not completed — Death | 41 | 26
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 2 | 8
Not completed — Sponsor decision | 1 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - AL101 4mg | Cohort 2 - AL101 6mg | Total
Number analyzed (Participants) | 45 | 42 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 27 | 62
  >=65 years | 10 | 15 | 25
Age, Continuous [Median (Full Range); unit: Years] | 50 [25 to 79] | 59 [25 to 80] | 56 [25 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 18 | 43
  Male | 20 | 24 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 31 | 33 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 6 | 14
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 1 | 4
  Netherlands | 0 | 4 | 4
  United States | 38 | 23 | 61
  United Kingdom | 3 | 5 | 8
  Israel | 0 | 3 | 3
  France | 1 | 3 | 4
  Spain | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as partial response (PR) + complete response (CR) as assessed by the investigator based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 for target lesions assessed by MRI.
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: 3 years and 7 months
Population: Efficacy evaluable analysis set includes all subjects who receive at least one complete infusion of study drug, have measurable disease at baseline per RECIST v1.1 or modified MDA criteria for bone-exclusive disease and have at least one post-baseline on-study assessment of tumor response.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - AL101 4mg | Cohort 2 - AL101 6mg
Number analyzed (Participants) | 41 | 36
Participants | 3 | 2

2. Secondary Outcome: Clinical Benefit Response Rate (CBR)
Description: Clinical benefit response rate (CBR) is defined as complete response (CR) + partial response (PR) + stable disease (SD) by investigator review based on RECIST v1.1 for target lesions assessed by MRI.
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Stable Disease (SD): Neither sufficient shrinkage (at least 30%) to qualify for PR nor sufficient increase (more than 20%) to qualify for PD, taking as reference the smallest sum diameters.
Time Frame: 3 years and 7 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - AL101 4mg | Cohort 2 - AL101 6mg
Number analyzed (Participants) | 41 | 36
Participants | 28 | 24

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined at the time from first infusion of investigational product to death due to any cause. Subjects with no documentation of death were censored at the last known date known to be alive.
Time Frame: 3 years and 5 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 - AL101 4mg | Cohort 2 - AL101 6mg
Number analyzed (Participants) | 41 | 36
months | 9.3 [6.6 to 14.2] | 9.4 [5.9 to 11.9]

ADVERSE EVENTS:
Time Frame: 3 years and 7 months
Description: The analysis was done on the safety population which consists of 87 patients (45 patients in the 4mg arm, and 42 patients in the 6mg arm) Safety analysis set includes all subjects who receive at least one infusion of study drug, including partial infusions..
Groups:
- Cohort 2 - AL101 6mg: AL101 6 mg mg once weekly (QW) intravenously (IV)
Arm/Group | Cohort 1 - AL101 4mg | Cohort 2 - AL101 6mg
All-Cause Mortality (participants affected / at risk) | 41/45 | 26/42
Serious Adverse Events (participants affected / at risk) | 23/45 | 26/42
Other Adverse Events (participants affected / at risk) | 45/45 | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - AL101 4mg (N=45) | Cohort 2 - AL101 6mg (N=42)
Pneumonia (Infections and infestations) | 4 | 2
Sepsis (Infections and infestations) | 2 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 1
Anorectal infection (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Brain abscess (Infections and infestations) | 1 | 0
Campylobacter sepsis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Cellulitis orbital (Infections and infestations) | 1 | 0
Meningitis bacterial (Infections and infestations) | 1 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 4
Dysphagia (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1
Ejection fraction decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Hepatobiliary disease (Hepatobiliary disorders) | 0 | 1
Bone marrow infiltration (Blood and lymphatic system disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Vasculitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - AL101 4mg (N=45) | Cohort 2 - AL101 6mg (N=42)
Diarrhoea (Gastrointestinal disorders) | 31 | 33
Nausea (Gastrointestinal disorders) | 30 | 19
Vomiting (Gastrointestinal disorders) | 21 | 13
Constipation (Gastrointestinal disorders) | 10 | 10
Dry mouth (Gastrointestinal disorders) | 7 | 13
Stomatitis (Gastrointestinal disorders) | 3 | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 3
Oral pain (Gastrointestinal disorders) | 3 | 4
Abdominal pain (Gastrointestinal disorders) | 5 | 1
Dysphagia (Gastrointestinal disorders) | 3 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 16
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Fatigue (General disorders) | 30 | 25
Asthenia (General disorders) | 2 | 7
Mucosal inflammation (General disorders) | 1 | 5
Pyrexia (General disorders) | 3 | 3
Chills (General disorders) | 3 | 1
Oedema peripheral (General disorders) | 1 | 3
Facial pain (General disorders) | 0 | 3
Swelling face (General disorders) | 0 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 25 | 18
Decreased appetite (Metabolism and nutrition disorders) | 10 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 5
Dehydration (Metabolism and nutrition disorders) | 2 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 7
Rash (Skin and subcutaneous tissue disorders) | 8 | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 7
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 5
Skin lesion (Skin and subcutaneous tissue disorders) | 6 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 3
Erythema (Skin and subcutaneous tissue disorders) | 1 | 3
Hair colour changes (Skin and subcutaneous tissue disorders) | 3 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 3
Headache (Nervous system disorders) | 13 | 4
Dysgeusia (Nervous system disorders) | 7 | 9
Dizziness (Nervous system disorders) | 6 | 4
Neuralgia (Nervous system disorders) | 0 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 0
Taste disorder (Nervous system disorders) | 3 | 0
Pneumonia (Infections and infestations) | 6 | 4
Urinary tract infection (Infections and infestations) | 3 | 3
Rash pustular (Infections and infestations) | 5 | 0
Oral candidiasis (Infections and infestations) | 1 | 3
Candida infection (Infections and infestations) | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Weight decreased (Investigations) | 7 | 11
Aspartate aminotransferase increased (Investigations) | 5 | 4
Alanine aminotransferase increased (Investigations) | 4 | 4
Platelet count decreased (Investigations) | 1 | 4
Neutrophil count increased (Investigations) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0
Insomnia (Psychiatric disorders) | 10 | 12
Anxiety (Psychiatric disorders) | 3 | 2
Depression (Psychiatric disorders) | 3 | 2
Vision blurred (Eye disorders) | 8 | 3
Dry eye (Eye disorders) | 1 | 4
Photophobia (Eye disorders) | 3 | 0
Hypertension (Vascular disorders) | 7 | 4
Infusion related reaction (Injury, poisoning and procedural complications) | 5 | 3
Anaemia (Blood and lymphatic system disorders) | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT03691207/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT03691207/SAP_001.pdf